CLINICAL TRIAL: NCT05785910
Title: Harmonization and Updating of Cognitive and Behavioral Assessment Procedures in Neurology: Adaptation of the Uniform Data Set for Telematic Administration
Brief Title: Adaptation of the Uniform Data Set for Telematic Administration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4074
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dementia, Mild; Dementia of Alzheimer Type
MeSH Terms: conditions — Dementia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal subjects (Experimental)
  Interventions: Diagnostic Test: IUDS

INTERVENTIONS:
Diagnostic Test: IUDS — a battery of neuropsychological test

SUMMARY:
The present project is an evolution of the previous RIN 2019 study aimed at validating and standardizing the Uniform Data Set (UDS) for dementia, a battery of tests exploring various cognitive domains (memory, language, praxis, executive functions) and involving partial tablet-based computerization for data collection.

In the present study, a UDS-based instrument that can be used in remote examiner-assisted telematic administration will be validated. This will be followed by standardization of the same on a sample of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* female and male subject between 50 and 90 years
* no negative score on the Anamnestic Questionnaire
* internist pathology in pharmacological compensation
* signing of informed consent

Exclusion Criteria:

* neurological pathologies
* decompensated metabolic pathology
* use of Benzodiazepine and psychoactive drugs

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
concordance index | from baseline through study completion, an average of 1 year and a half
  Measure the concordance index in the administration of individual battery tests between in-person and computer-based administration

SECONDARY OUTCOMES:
regression lines | from baseline through study completion, an average of 1 year and a half
  Describe for each individual test the regression lines and correction factors for the interfering demographic variables (age schooling and sex)

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Marra, MD, Principal Investigator — Memory clinic, Fondazione Policlinico Gemelli, IRCCS, Università Cattolica del Sacro Cuore
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Clinica della memoria, Rome, Lazio, Italy